CLINICAL TRIAL: NCT02459951
Title: Improving Holding Function of the Hemiplegic Hand With Chemodenervation
Brief Title: Improving Holding Function of the Hemiplegic Hand
Status: Completed | Type: Observational
Sponsor: Nathaniel Mayer (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Nathaniel Mayer, Director, Motor Control Analysis Laboratory MossRehab, Albert Einstein Healthcare Network
Organization: Albert Einstein Healthcare Network (Other)
Other Study IDs: 4729FBD
Record Dates: First submitted 2015-05-14; First posted 2015-06-02 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: Muscle Spasticity; Botox A; Upper limb hemiplegia
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- clenched fist: Adult participants with upper limb hemiparesis secondary to stroke and greater than 12 months duration. Medical determination that .botulinum toxin injections are indicated for treatment of spasticity.
  Interventions: Other: clenched fist

INTERVENTIONS:
Other: clenched fist — Observation of performance on a standardized behavioral task pre- and post- administration of Botox A in the context of routine care. Clinical assessment and judgment will be used to determine dosing and which muscles contribute to the hand deformities of a given participant.

SUMMARY:
Relevant to patients with spastic hemiparesis in the hand and upper limb, this pilot project proposes to measure the effects of botulinum toxin injections through observation of performance on a functional task known as 'hand as a holder'. This task requires the person with hemiplegia to insert an object into the affected hand and hold it independently.

The project aims to demonstrate reliability and validity of a digital video method that will be used to measure 'insertion time'. It also aims to establish initial statistical support for improved object insertion time into the hemiplegic clenched fist after Botox A injections.

DETAILED DESCRIPTION:
Holding is an everyday hand function, objects entering the hand radially, frontally, ulnarly or in-between the finger spaces. After a stroke, the hand of a person with hemiplegia typically lacks voluntary finger extension that opens the hand. Simultaneously, the hand is also subjected to involuntary contraction of finger flexor muscles that close the hand, resulting in clenched fist and thumb-in-palm deformities. Despite these typical hemiplegic configurations, persons with stroke may be able to insert an object into the hand by wiggling and pushing it into the hemiplegic hand with their uninvolved hand, though struggle is often present and failure is frequent. In the hemiplegic patient, a common driver of clenched fist and thumb-in-palm configurations is excessive involuntary neural activation of finger and thumb flexors, compounded by impaired or absent voluntary finger extension. Excessive finger and thumb flexor contractions have been variously ascribed to involuntary phenomena such as spasticity, spastic dystonia, co-contraction, associated reactions and others. For the investigators purpose here, these involuntary phenomena generate contractile tension in hand and thumb muscles that choke the hand's potential to function as a holder of objects as described above.

The underlying rationale of this project is to examine whether hemiplegic 'hand as a holder' function can be improved by weakening involuntary muscle contractions that generate clenched fist and thumb in palm using the neuromuscular blocking properties of Botox A. The investigators hypothesize that 'hand as a holder' function will improve after chemodenervation of relevant finger, thumb and wrist muscles selected by clinical examination.

Nine subjects will be enrolled. Baseline observations will be made on two occasions prior to Botox A injection and outcomes measured four weeks later. A digital video method will be used to measure 'insertion time' at all-time points. Given the importance of the relationship between "statistically significant" research results and "clinically significant", person-oriented, functional improvement, the investigators also hypothesize that experienced clinicians will independently rate the performance of object insertion into the clenched fist as globally better after chemodenervation.

ELIGIBILITY:
Inclusion Criteria:

* patients who are clinically appropriate for treatment of upper limb spasticity due to stroke with Botox A injections ;
* adults up to age 80, women must be post-menopausal or are medically unable to conceive (as determined from their medical records), men must be at least age 35
* documented anemic or hemorrhagic unilateral (right or left) hemiplegic stroke, with 1 year or more prior to enrollment
* able to understand verbal and visual instructions and demonstrations regarding the protocol
* a resting wrist angle equal to or less than 0
* spasticity is present in finger flexors and thumb coupled with marked voluntary paresis of finger extension (no finger has more than half range of active extension at any joint). By squeezing the examiner's finger, participants will have demonstrated, at least, some detectable voluntary contraction of finger flexors; impaired sensation is acceptable but participants must be aware that they are holding something, as tested clinically;
* at least two finger flexors with an Ashworth score = 3;
* moderate motor severity as defined by an upper limb Fugl-Meyer motor scores between 21-50
* normal joint capsule without contractures as determined by clinical exam; participant may have tightness/shortening of extrinsic finger flexors but composite extension of wrist and fingers comes to at least neutral (i.e. fingers and wrist can be brought to neutral position simultaneously).

Exclusion Criteria:

* profound sensory loss/absent touch sensation
* known hypersensitivity/allergy to Botox A
* acute illness or unresolved medical/psychiatric conditions at time of assessment
* symptomatic lung disease and compromised respiratory status; muscle-weakening neurological disorders known to increase drug-related risk [e.g. amyotrophic lateral sclerosis (ALS), myasthenia gravis, Lambert-Eaton syndrome, or motor neuropathy]
* infection in the area where the study drug should be injected
* pregnancy or breast-feeding;
* participant had Botox injections less than 4 months previously
* clenched fist associated with tenodesis of an extended wrist i.e. resting position of wrist is > 0 degrees

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are clinically appropriate for Botox A injection to treat upper limb spasticity due to stroke
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Mayer, MD, Principal Investigator — Albert Einstein Healthcare Network

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer NH, Ferraro M, Pauloski-Hunt D, Chervoneva I. Capacity for Hand-as-a-Holder Function of the Spastic Combination Hand: A Proof-of-Concept Study. Am J Phys Med Rehabil. 2022 Mar 1;101(3):298-302. doi: 10.1097/PHM.0000000000001834. PMID 34173778

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemiplegic Clenched Fist: Adult participants with upper limb hemiparesis secondary to stroke and greater than 12 months duration. Medical determination that .botulinum toxin injections are indicated for treatment of spasticity.
  clenched fist: Observation of performance on a standardized behavioral task pre- and post- administration of Botox A in the context of routine care. Clinical assessment and judgment will be used to determine dosing and which muscles contribute to the hand deformities of a given participant.
Period: Overall Study
Arm/Group | Hemiplegic Clenched Fist
Started | 10
Completed | 9
Not Completed | 1
Not completed — Unable to meet holding requirement | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hemiplegic Clenched Fist
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 61 [52 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9
Months post stroke [Mean (Full Range); unit: months] | 64 [24 to 102]
Fugl-Meyer Assessment (upper limb motor score only) [Mean (Full Range); unit: units on a scale] — Scale range is 0 to 66 (upper extremity motor score only); higher score is better
  units on a scale | 24 [10 to 47]
Weinstein Enhanced Sensory Test (West) [Mean (Full Range); unit: units on a scale] — scale measures sensation using monofilament pressure; scale range is: 1.65 -6.65; lower score is better
  units on a scale | 4.42 [2.83 to 6.65]
Visual Neglect [Count of Participants; unit: Participants] — The presence of visual neglect as determined by clinical examination
  Participants | 0
dominant hand is affected [Count of Participants; unit: Participants] | 4
days between the two baseline evaluations [Mean (Full Range); unit: days] | 6 [2 to 14]
days post injection evaluation [Mean (Full Range); unit: days] — number of days after participants were injected with OnabotulinumtoxinA and then evaluated
  days | 26 [21 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Geometric Ratios of Log-transformed Transit Time
Description: Time (log-transformed) required for contralateral hand to insert a plastic cylinder successfully into the hemiplegic clenched fist AND assessed at Pre-injection baseline 2 and a Post-injection session expressed as a geometric mean ratio of these sessions. (Success is defined by a hold of 5 secs or more). Geometric mean ratios are calculated for each of 5 cylinder sizes (A-E)
Time Frame: days post-injection evaluation (mean 26 days; range 21-30 days)
Measure: Geometric Mean (95% Confidence Interval); unit: dimensionless ratio
Arm/Group | Hemiplegic Clenched Fist
Number analyzed (Participants) | 9
dimensionless ratio
  cylinder A (.5 " diameter) | 1.19 [0.99 to 1.41]
  cylinder B (1" diameter) | 1.07 [0.89 to 1.27]
  cylinder C (1.5" diameter) | 0.79 [0.65 to 0.97]
  cylinder D (2" diameter) | 0.72 [0.57 to 0.90]
  cylinder E (2.5" diameter) | 0.66 [0.51 to 0.85]
Statistical Analysis 1: Comparison: Hemiplegic Clenched Fist; Test type: Superiority; p = .059, Regression, Logistic — refer to cylinder A (.5" diameter)
Statistical Analysis 2: Comparison: Hemiplegic Clenched Fist; Test type: Superiority; p = 0.465, Regression, Logistic; refer to cylinder B(1" diameter); geometric mean ratio B
Statistical Analysis 3: Comparison: Hemiplegic Clenched Fist; Test type: Superiority; p = .022, Regression, Logistic — refer to cylinder C (1.5" diameter); geometric mean ratio C
Statistical Analysis 4: Comparison: Hemiplegic Clenched Fist; Test type: Superiority; p = .004, Regression, Logistic — refer to cylinder D (2" diameter); geometric mean ratio D
Statistical Analysis 5: Comparison: Hemiplegic Clenched Fist; Test type: Superiority; p = .002, Regression, Logistic — refer to cylinder E (2.5" diameter); geometric mean ratio E

2. Secondary Outcome: Fraction of Successful Holds for Each Evaluation Session
Description: fraction of successful holds for each evaluation session (Pre1, Pre2, and Post)
Time Frame: days between two baseline evaluations (mean 6; range 2-14) and days post-injection evaluation (mean 26; range 21-30)
Measure: Mean (95% Confidence Interval); unit: fraction of successful holds
Arm/Group | Hemiplegic Clenched Fist
Number analyzed (Participants) | 9
fraction of successful holds
  post injection | .67 [.48 to .95]
  pre 1 baseline | .51 [.37 to .72]
  pre2 baseline | .53 [.37 to .77]

3. Secondary Outcome: Ratio of Successful Holds
Description: ratio of successful holds post/pre1, post/pre2 or pre1/pre2
Time Frame: days between two baseline evaluations (mean 6; range 2-14) and days post-injection evaluation (mean 26; range 21-30)
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Clenched Fist
Number analyzed (Participants) | 9
ratio
  post vs. pre1 | 1.31 [1.05 to 1.64]
  post vs pre2 | 1.26 [1.02 to 1.57]
  pre1 vs pre2 | .96 [.71 to 1.3]

4. Other Pre Specified Outcome: Modified Ashworth Score (MAS)
Description: A clinical ordinal measure of resistance to passive stretch of a limb on a scale of 0-4 with higher scores representing greater resistance
Time Frame: days between two baseline evaluations (mean 6; range 2-14) and days post-injection evaluation (mean 26; range 21-30)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Clenched Fist
Number analyzed (Participants) | 9
units on a scale
  Pre2 vs Pre1 | 0 [0 to 1.5]
  Post vs. Pre1 | -2 [-2 to -1.5]
  Post vs. Pre2 | -2 [-2 to -1.5]

ADVERSE EVENTS:
Time Frame: until 5 weeks post injection
Arm/Group | Hemiplegic Clenched Fist
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02459951/Prot_SAP_000.pdf